CLINICAL TRIAL: NCT01338090
Title: 89Zr-bevacizumab PET Imaging as Predictive Biomarker for Everolimus Efficacy in Patients With Neuroendocrine Tumors
Brief Title: 89Zr-bevacizumab PET Imaging in Patients With Neuroendocrine Tumors
Acronym: NETPET
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Prof.dr. E.G.E. de Vries, University Medical Center Groningen
Other Study IDs: 20091104; 2009-017195-24 (EudraCT Number)
Record Dates: First submitted 2011-04-12; First posted 2011-04-19 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2011-08

CONDITIONS: Neuroendocrine Tumors
Keywords: VEGF imaging; neuroendocrine tumors; biomarker; mTOR inhibition
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 89Zr-bevacizumab; Everolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 89Zr-bevacizumab
  Interventions: Drug: 89Zr-bevacizumab; Drug: Everolimus

INTERVENTIONS:
Drug: 89Zr-bevacizumab — Intravenous injection 120 MBq
Drug: Everolimus — Oral use, 10 mg per day
  Other Names: RAD001

SUMMARY:
This is a pilot study for evaluation of 89Zr-bevacizumab PET imaging as predictive biomarker during treatment with everolimus in patients with neuroendocrine tumors.

Patients with progressive disease during the last year will receive treatment with everolimus 10 mg/day orally and 89Zr-bevacizumab PET imaging will be performed before start of treatment and after 2 and 12 weeks of treatment in the first three patients. If the scan after 2 weeks of treatment is already informative further patients will not undergo a scan at 12 weeks. A scan is considered already informative if both scans show at least 30% decrease in uptake in case of response, or at least 30% increase in uptake in case of disease progression.

Four days before the scan patients will be injected intravenously 37 MBq, protein dose 5 mg 89Zr-bevacizumab. At day 1, day 15 and day 99, PET images will be made for visualization and quantification of VEGF in the tumor lesions and blood will be drawn for determination of angiogenesis and mTOR pathway related biomarkers.

DETAILED DESCRIPTION:
1. Rationale:

   Profound angiogenesis is an important characteristic of neuroendocrine tumors. Antiangiogenic drugs including sunitinib, bevacizumab and everolimus have shown antitumor activity in neuroendocrine tumors. The investigators participated in the RAD001 studies for neuroendocrine tumors. From preclinical studies including studies performed in our own lab the investigators know that everolimus downregulates VEGF.

   Currently it is not possible to predict which individual patient will benefit from treatment with an mTOR inhibitor. A predictive biomarker for efficacy of mTOR inhibitors is urgently needed and would be helpful, as a predictive biomarker may facilitate the development of combination therapies, of individual titration of the dose, and it may facilitate early clinical studies. Furthermore, it may spare the patients unnecessary side effects. mTOR inhibitors may fail in individual patients because angiogenesis is not sufficiently inhibited. Non-invasive imaging of VEGF before and early after start of treatment may have predictive value for treatment efficacy.

   Within the UMCG the investigators have an active ongoing research line on molecular imaging. The investigators have developed as part of this the 89Zr-bevacizumab PET label for non-invasive measurement of VEGF levels in the tumor and its surrounding microenvironment. This tracer can give insight in the tumors' dependency on angiogenesis as the investigators have already proven for a VEGF-receptor tyrosine kinase inhibitor. Currently this tracer is used in clinical trials. The investigators would like to examine whether all neuroendocrine tumors produce VEGF and whether they differ in their response to inhibition of VEGF by mTOR.
2. Objectives:

The primary objective is to evaluate the feasibility of 89Zr-bevacizumab-PET imaging as predictive biomarker before and during treatment with everolimus in patients with neuroendocrine tumors.

The secondary Objectives are the following:

* To explore if 89Zr-bevacizumab PET imaging can differentiate patients with progressive neuroendocrine tumors from patients with non-progressive disease early during treatment with everolimus.
* To explore relationships between VEGF pathway related blood biomarkers and changes in 89Zr-bevacizumab tumor uptake.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with metastatic neuroendocrine tumors
* radiological documentation of progressive disease over the past year
* measurable disease according to RECIST criteria
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb > 9 g/dL.
* Adequate liver function: serum bilirubin: ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN. Patients with known liver metastases: AST and ALT ≤ 5x ULN.
* Adequate renal function: serum creatinine ≤ 1.5 x ULN.
* Fasting serum cholesterol ≤300 mg/dL OR 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In cases where one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication

Exclusion Criteria:

* uncontrolled medical conditions (eg, unstable angina, symptomatic heart failure, serious intercurrent infections)
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule of the study
* Patients with uncontrolled diabetes mellitus as defined by fast blood sugar > 1.5 x ULN.
* Prior therapy with RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus).
* Concomitant medications known to inhibit, induce or be a substrate to isoenzyme CYP3A are excluded unless the drugs are medically necessary and no substitutes are available. If there are no acceptable substitutes, special precautions should be taken in these patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic neuroendocrine tumors.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change in 89Zr-bevacizumab uptake | 12 weeks
  The change in 89Zr-bevacizumab uptake in tumor lesions between the baseline PET scan and the scans performed after 2 and 12 weeks of everolimus treatment in patients with neuroendocrine tumors. In addition, effect sizes and confidence intervals will be determined.

SECONDARY OUTCOMES:
Progressive disease | 12 weeks
  Progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST)22 criteria on CT after 12 weeks of treatment.
  Progression is defined as the appearance of new disease or an increase of 20% in the sum of the longest diameters of the target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth GE de Vries, MD, PHD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands